CLINICAL TRIAL: NCT02045225
Title: An HIV Prevention Intervention for HIV-negative Men Who Have Sex With Men Via Reduction of Social Anxiety and Substance Use in Sexual Situations
Brief Title: HIV Prevention for HIV-Negative Men Via Reduction of Social Anxiety
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Trevor Hart, Principal Investigator, Toronto Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201203HHP-279414-PB1ABAF146056; 201203HHP-279414 (Other: CIHR)
Record Dates: First submitted 2013-05-24; First posted 2014-01-24 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Social Anxiety; Substance Use
Keywords: social anxiety in sexual situations
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive behavioural therapy (Experimental): Reduction of social anxiety & substance use in gay/bi men
  Interventions: Behavioral: Reduction of social anxiety & substance use in gay/bi men

INTERVENTIONS:
Behavioral: Reduction of social anxiety & substance use in gay/bi men — The study will provide Phase I trial data for a novel and innovative HIV prevention intervention for MSM built upon empirically supported interventions to reduce HIV risk among MSM and cognitive-behavioural therapy to reduce social anxiety. This study will test a novel integrated HIV prevention intervention that combines empirically supported treatments for social anxiety with HIV risk reduction counseling to reduce HIV sexual risk behaviour. Study objectives: 1) to provide data on the acceptability/feasibility of the intervention, 2) to provide data to test the intervention, and 3) to provide data that will allow for a RCT that will test intervention efficacy relative to HIV prevention interventions that do not reduce social anxiety or substance use in sexual situations.

SUMMARY:
Men who have sex with men (MSM) bear a disproportionate burden of the Human Immunodeficiency Virus (HIV) epidemic in Canada, and HIV incidence appears to be rising among Canadian MSM (1). MSM comprised nearly half (44.1%) of new positive HIV tests in 2009 (2). Among MSM in Ontario, from 2001 to 2006, HIV diagnoses increased 26% (3). Given the alarmingly high HIV prevalence rates among MSM in North American cities, there is a critical need for HIV prevention interventions for MSM in Canada. Social anxiety, or anxiety about being evaluated in interpersonal situations, is a reliable risk factor for unprotected anal intercourse (UAI) among MSM (4 and 5). Social anxiety is highly modifiable via cognitive-behavioural therapy, a form of psychotherapy (6). Social anxiety may also increase substance use in sexual situations, which is another risk factor for HIV among MSM (7 and 8). As such, an empirically-based social anxiety treatment may also reduce HIV risk behaviours among MSM. The present study will provide Phase I trial data for a novel and innovative HIV prevention intervention for MSM. This is a proposal to test a novel integrated HIV prevention intervention that combines empirically supported treatments for social anxiety with HIV risk reduction counseling to reduce HIV sexual risk behaviour.

DETAILED DESCRIPTION:
The present study will provide pilot data for a novel and innovative HIV prevention intervention for MSM. This intervention will build upon empirically supported interventions to reduce HIV risk among MSM and cognitive-behavioural therapy to reduce social anxiety. This pilot study will serve 3 related major objectives: 1) to provide data on the acceptability and feasibility of the intervention administered, 2) to provide pilot data testing the intervention, and 3) to provide data that will allow Dr. Hart and his team to apply to CIHR for a Phase II trial that will test the efficacy of the intervention relative to HIV prevention interventions that do not reduce social anxiety or substance use in sexual situations among MSM.

Participants attend 4 assessment sessions, during which they complete a series of interviews and questionnaires regarding social anxiety, substance use, and sexual risk behaviours. Participants also attend 10 sessions of counselling, where a therapist seeks to help the participant work towards reducing his anxiety in social and sexual situations and try to better manage his use of alcohol and drugs in sexual situations. The participant undergoes a baseline assessment, followed by 10 weekly counselling sessions, a post-treatment assessment, and 3- and 6-month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years
* male identified
* gay or bisexual identified
* experiencing social anxiety in sexual situations
* condomless anal sex with a casual (or non-monogamous) HIV-positive or unknown serostatus partner in the last 3 months
* consumption of alcohol and/or a recreational drug within 2 hours before sex or during sex within the last 3 months

Exclusion Criteria:

* younger than 18 or older than 65 years of age
* not male identified
* sexual orientation other than gay or bisexual
* no experiences of social anxiety in sexual situations
* severe mental illness
* already receiving psychotherapy

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Instances of unprotected anal intercourse with sexual partners who are HIV-positive or of unknown HIV status | 3, 6, and 9 months following baseline assessment
  Sexual Behavior and Related Measures:
  Sexual Risk Behavior and Related Assessment (self-report)

SECONDARY OUTCOMES:
Severity of social anxiety and instances substance use in sexual situations | 3, 6, and 9 months after baseline assessment
  Social Anxiety Measures:
  Social Interaction Anxiety Scale (SIAS) Social Phobia Scale (SPS) Liebowitz Social Anxiety Scale (LSAS) Anxiety Disorders Interview Schedule (ADIS-DSM-IV) Brief Fear of Negative Evaluation Scale, Straightforward Items (BFNE-S)
  Substance Use Measures:
  The Alcohol Use Disorders Identification Test (AUDIT) Brief Michigan Alcohol Screening Test (BMAST) The Addictions Severity Index Lite (ASI-Lite)

CONTACTS AND LOCATIONS:
Overall Officials: Trevor A Hart, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Ryerson University, Toronto, Ontario, Canada

REFERENCES:
- [Background] Remis RS, Swantee C, Schiedel L, Liu J. Report on HIV/AIDS in Ontario. March, 2008. http://www.health.gov.on.ca/english/providers/pub/aids/reports/report_hivaids_ontario_2006.pdf.
- [Background] Public Health Agency of Canada. (2010). HIV and AIDS in Canada: Surveillance report to December 31, 2009. http://www.phac-aspc.gc.ca/aids-sida/publication/index-eng.php#surveillance.
- [Background] Hart TA, Heimberg RG. Social anxiety as a risk factor for unprotected intercourse among gay and bisexual male youth. AIDS Behav. 2005 Dec;9(4):505-12. doi: 10.1007/s10461-005-9021-2. PMID 16205961
- [Background] Hart TA, James CA, Purcell DW, Farber E. Social anxiety and HIV transmission risk among HIV-seropositive male patients. AIDS Patient Care STDS. 2008 Nov;22(11):879-86. doi: 10.1089/apc.2008.0085. PMID 19025482
- [Background] Hofmann SG, Smits JA. Cognitive-behavioral therapy for adult anxiety disorders: a meta-analysis of randomized placebo-controlled trials. J Clin Psychiatry. 2008 Apr;69(4):621-32. doi: 10.4088/jcp.v69n0415. PMID 18363421
- [Background] Semple SJ, Strathdee SA, Zians J, McQuaid J, Patterson TL. Psychosocial and behavioral correlates of anxiety symptoms in a sample of HIV-positive, methamphetamine-using men who have sex with men. AIDS Care. 2011 May;23(5):628-37. doi: 10.1080/09540121.2010.525608. PMID 21293993
- [Background] Elkington KS, Bauermeister JA, Zimmerman MA. Psychological distress, substance use, and HIV/STI risk behaviors among youth. J Youth Adolesc. 2010 May;39(5):514-27. doi: 10.1007/s10964-010-9524-7. Epub 2010 Mar 14. PMID 20229264